CLINICAL TRIAL: NCT06595134
Title: AI for the Prediction of Obesity-Related Vascular Diseases - Validation Study
Brief Title: AI-POD Clinical Validation Study for Obese Patients
Acronym: AI-POD
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Bonn (Other)
Collaborators: European Union (Other)
Responsible Party: Principal Investigator, Prof. Dr. Ulrike Attenberger, Director, Clinic for Diagnostik and Interventional Radiology, University Hospital, Bonn
Other Study IDs: 310/23-EP
Record Dates: First submitted 2024-05-13; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Acute Cardiovascular Disease
Keywords: Obesity, Heart CT, Artificial Intelligence
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Arm 1: Standard Care plus Fitnesstracker and Citizen App
  Interventions: Other: Non Interventional
- Arm 2: Standard Care
  Interventions: Other: Non Interventional

INTERVENTIONS:
Other: Non Interventional — Screening (Day -7 to Day -1) Visit 1 (Day 0) Visit 2 (Month 3 +/- 7 days) Visit 3 (Month 6 +/- 7 days) Visit 4 (Month 12 +/- 7 days) Visit 5 (Month 24 +/- 7 days) Visit 6 (Month 60 +/- 30 days; end of study)

SUMMARY:
The study is aimed at patients who suffer from severe obesity and receive a computerised tomography (CT) scan of the heart. A total of 1200 patients across Europe are to take part in the study. It is a multi-centre, controlled, open, randomised study. As part of the study, a citizen app will be installed on a smartphone for randomly selected study participants. A fitness tracker will also be issued so that certain parameters, such as heart rate and daily number of steps, can be recorded.

DETAILED DESCRIPTION:
The clinical validation study of the AI-POD instruments (risk score, CDSS, Citizen App) is designed as a prospective, multicentre observational study. Obese patients (BMI >30 kg/m2) with suspected CVD who are scheduled for a cardiac CT scan (consisting of calcium scoring and coronary CT angiography) will be included in the study. This clinically indicated cardiac CT scan will serve as a baseline examination, and a second cardiac CT scan will be performed after a follow-up period of 2 years. Both cardiac CT examinations will be performed on a photon-counting CT system (PCCT). In addition to the CT data, clinical data (anthropometry and physical parameters such as body weight, height, age, gender, BMI, waist circumference, waist-to-hip ratio, body impedance analysis, cardiovascular risk factors, medication, previous interventions and operations) will be collected, symptoms and results of echocardiography to determine left ventricular function) as well as laboratory data on (subclinical) inflammation (hsCRP, leukocytes, monocyte activation), lipid disorders (HDL, LDL, total cholesterol, triacylglycerides), glucose homeostasis (HbA1c, fasting glucose, HOMA index), liver and kidney function (creatinine, GFR, GOT/ALAT, GPT/ASAT) are collected at a total of 5 visits over 2 years. Half of all included patients will also be randomised to receive access to the Citizen app and a separate fitness tracker device to record the following data: Activity data such as step count, heart rate, height, weight, gender, age, waist circumference circumference, nutritional data such as calorie intake, nicotine, alcohol, sleep.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 45 years at the time of signing informed consent
* BMI greater than or equal to 30 kg/m2
* Patients with suspected CVD (>15% pretest probability [ESC guidelines]), referred for cardiac CT examinations (consisting of coronary calcium scoring and coronary CT angiography)
* Informed consent of the patient

Exclusion Criteria:

* Any of the following CV conditions within 2 months prior to study inclusion: myocardial infarction, stroke,
* Hospitalization for unstable angina pectoris or transient ischemic attack or due to congestive heart failure.
* Planned coronary, carotid, or peripheral artery revascularisation known on the day of inclusion
* Presently classified NYHA IV heart failure
* Having uncontrolled diabetes mellitus (HbA1c ≥ 11%) at day of inclusion
* Having uncontrolled hypertension (SBP ≥ 160 mmHg and/or DBP ≥ 100 mmHg) as measured at inclusion
* Having severe renal impairment measured as an eGFR < 30 mL/min/1.73 m2 at inclusion
* Alanine aminotransferase (ALT) or alkaline phosphatase (APT) level < 3.0 x the upper limit of normal (ULN)for the reference range
* Total bilirubin level >1.5 x the ULN for the reference range
* History of an active or untreated malignancy or are in remission from a clinically significant malignancy for less than 5 years
* Previous organ transplantation or awaiting an organ transplant
* Pregnancy or breastfeeding

Min Age: 45 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Obese patients (BMI >30 kg/m2) with suspected CVD and scheduled for a cardiac CT examination (consisting of calcium scoring and coronary CT angiography).
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
An improved accuracy in prediction of CVD progression by us-ing the AI-POD risk score | Between Visit 1 and Visit 5 (Day 0 and Month 24)
  Change in plaque volume
An improved accuracy in prediction of CVD progression by us-ing the AI-POD risk score | Between Visit 1 and Visit 5 (Day 0 and Month 24)
  Change in plaque com-position/CAC
An improved accuracy in prediction of CVD progression by us-ing the AI-POD risk score | Between Visit 1 and Visit 5 (Day 0 and Month 24)
  Change in luminal stenosis

SECONDARY OUTCOMES:
To validate the Citizen App, to assess the improvement of AI-POD risk score Accuracy and feasibility of collecting data with citizen App | After 2 Years
  Time-to-first occurrence of HbA1c greater than or equal to 48 mmol/mol (6.5%) for subjects with screening HbA1c < 6.5 mmol/mol at study inclusion
To validate the Citizen App, to assess the improvement of AI-POD risk score Accuracy and feasibility of collecting data with citizen App | After 2 Years
  Change in systolic blood pressure (mmHg)
To validate the Citizen App, to assess the improvement of AI-POD risk score Accuracy and feasibility of collecting data with citizen App | After 2 Years
  Change in diastolic blood pressure (mmHg)
To validate the Citizen App, to assess the improvement of AI-POD risk score Accuracy and feasibility of collecting data with citizen App | After 2 Years
  Change in pulse rate
To validate the Citizen App, to assess the improvement of AI-POD risk score Accuracy and feasibility of collecting data with citizen App | After 2 Years
  Change in body weight (Kgs)
To validate the Citizen App, to assess the improvement of AI-POD risk score Accuracy and feasibility of collecting data with citizen App | After 2 Years
  Change in fat mass (BIA); weight and height will be combined to report BMI in kg/m^2
To validate the Citizen App, to assess the improvement of AI-POD risk score Accuracy and feasibility of collecting data with citizen App | After 2 Years
  Change in waist circumference (cm)
To validate the Citizen App, to assess the improvement of AI-POD risk score Accuracy and feasibility of collecting data with citizen App | After 2 Years
  Change in HbA1c
To validate the Citizen App, to assess the improvement of AI-POD risk score Accuracy and feasibility of collecting data with citizen App | After 2 Years
  Change in total cholesterol, LDL, HDL, hsCRP, transaminases
To validate the Citizen App, to assess the improvement of AI-POD risk score Accuracy and feasibility of collecting data with citizen App | After 2 Years
  MACE (Major Adverse Cardiac Event)

CONTACTS AND LOCATIONS:
Overall Officials: Ulrike Attenberger, Prof. Dr., Principal Investigator — ulrike.attenberger@meduniwien.ac.at
Locations (6):
- Medical University Vienna, Vienna, Austria
- University Hospital Leuven, Leuven, Belgium
- University Hospital Pilsen, Pilsen, Czechia
- Germany (2):
  - University Hospital Bonn, Bonn, North Rhine-Westphalia
  - University Hospital Mannheim, Mannheim
- University Hospital Zürich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided